CLINICAL TRIAL: NCT06436391
Title: Effect of Kinesio Tape and ShotBlocker on Pain, Comfort and Crying Duration in Heel Blood Collection in Infants: Randomized Controlled Trial
Brief Title: The Effectiveness of Two Different Methods in Heel Blood Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: Selcuk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: He1
Record Dates: First submitted 2024-05-08; First posted 2024-05-31 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Infant Behavior; Pain
Keywords: Pain Management; Kinesiotape; Nursing; Therapy
MeSH Terms: conditions — Infant Behavior; Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: The study will be conducted with infants of mothers who meet the inclusion criteria and agree to participate in the study. After explaining the study to the parents, the study will start after obtaining their verbal and written consent. Randomization will be random assignment to a control group or two intervention groups (1:1:1) with sequentially numbered, sealed, opaque envelopes containing randomly generated numbers after mothers have obtained informed consent. Randomization will be carried out via www.random.org using a table of random numbers. This will be done by an independent statistician and envelopes will be given to the researchers
Who Masked: Participant
Masking Description: Single Blinded for mothers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio tape group (Experimental): To the infants in the experimental group; Kinesio tape application will be performed by an experienced physiotherapist whom has a M.Sc. degree and kinesio tape certificate.
  Interventions: Other: Kinesio taping
- ShotBlocker group (Experimental): To the infants in the second experimental group; Shotblocker application will be performed by another researcher.
  Interventions: Other: ShotBlocker
- Control group (No Intervention): These infants will not receive any intervention in the heel prick procedure. Routine heel blood collection will be performed.

INTERVENTIONS:
Other: Kinesio taping — Kinesio taping will be applied to the lateral part of the baby's heel to increase blood flow. Blood collection will always be performed by the same nurse
  Arms: Kinesio tape group
Other: ShotBlocker — Shotblocker will be applied to the baby's heel average 10-15 seconds with minimal pressure.
  Arms: ShotBlocker group

SUMMARY:
This study aims to evaluate the effectiveness of 2 non-pharmacological methods that will reduce the traumatizing effect of routine heel pricking in infant babies within the scope of the metabolic endocrine screening program. One of the interventions to be used in the study is kinesio taping, a type of taping that does not contain any medication. Another intervention is Shotblocker, which does not belong to any drug or device group.

DETAILED DESCRIPTION:
Studies on pain indicate that severe pain experienced in the early period of life causes a weakening of the cognitive functions of the infant, especially by shrinking the thalamic volume. Pain management in the neonatal period aims to help the infant cope with pain by relieving it. For effective pain management, it is very important to diagnose and evaluate the baby's response to pain early and accurately within a multidisciplinary team approach, and to select appropriate interventions to alleviate the pain experience. It is stated that nonpharmacological methods in relieving procedural pain strengthen the baby's natural regulation and coping mechanisms when faced with painful intervention and reduce pain and stress. For this reason, this study aimed to determine the effect of kinesiology taping and ShotBlocker applied to the heel during heel blood collection in infant babies on pain, comfort and crying time.

ELIGIBILITY:
Inclusion Criteria:

* Term birth infants,
* Infants with a birth weight of 2500 g and above
* Infants with stable clinical condition
* Infants who can perform vital functions without support,
* Infants who were fed, calm and not crying within one hour before the procedure will be included.

Exclusion Criteria:

* With a genetic or congenital anomaly,
* Neurological, cardiological and metabolic diseases,
* In need of respiratory support,
* Infants receiving analgesics, antiepileptics before the procedure will be excluded.

Ages: 38 Weeks to 41 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Determining the descriptive characteristics of infants | Average 5 minutes
  1-Infant Introduction Form The questionnaire created by the researchers consisted of a total of 10 questions including infant gender, gestational age, postnatal age, birth weight and some demographic characteristics.
Follow-up of infants | Average 5 minutes
  2- Infant Follow-up Form: This form is the form to record the duration of the procedure and the duration of crying.
The effect of Kinesio tape and ShotBlocker on pain | Average 5 minutes
  3- Neonatal Infant Pain Scale (NIPS):This scale, which was developed in 1993 to evaluate behavioral and physiological pain responses of preterm and term infants, was adapted into Turkish in 1999. A high score indicates that the severity of pain.

SECONDARY OUTCOMES:
The effect of Kinesio tape and ShotBlocker application in infants in the experimental groups' comfort . | Average 5 minutes
  1-COMFORTneo scale: The scale was revised under the name COMFORTneo scale and its validity and reliability were established. COMFORTneo measures only behavioral parameters in the newborn without physiological parameters. It is Likert-type and evaluates the comfort needs, pain and distress of newborns followed up in intensive care. The lowest score that can be obtained from the scale is 6 and the highest score is 30. As the score increases, it is understood that the baby is not comfortable and needs interventions to provide comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel KUCUKOGLU, Ph.D., Principal Investigator — Selcuk University
Locations (1):
- Nigde Omer Halisdemir Eğitim ve Araştırma Hastanesi, Niğde, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published

REFERENCES:
- [Background] Chik YM, Ip WY, Choi KC. The Effect of Upper Limb Massage on Infants' Venipuncture Pain. Pain Manag Nurs. 2017 Feb;18(1):50-57. doi: 10.1016/j.pmn.2016.10.001. Epub 2016 Dec 10. PMID 27964912
- [Background] Anand KJ, Hickey PR. Pain and its effects in the human neonate and fetus. N Engl J Med. 1987 Nov 19;317(21):1321-9. doi: 10.1056/NEJM198711193172105. No abstract available. PMID 3317037
- [Background] Erkut Z, Yildiz S. The Effect of Swaddling on Pain, Vital Signs, and Crying Duration during Heel Lance in Newborns. Pain Manag Nurs. 2017 Oct;18(5):328-336. doi: 10.1016/j.pmn.2017.05.007. Epub 2017 Aug 2. PMID 28779961
- [Background] Foster JP, Taylor C, Spence K. Topical anaesthesia for needle-related pain in newborn infants. Cochrane Database Syst Rev. 2017 Feb 4;2(2):CD010331. doi: 10.1002/14651858.CD010331.pub2. PMID 28160271
- [Background] Harvey EG. Kinesio taping to address post-sternotomy scars in pediatric patients: A case report. Scars Burn Heal. 2022 May 11;8:20595131221095355. doi: 10.1177/20595131221095355. eCollection 2022 Jan-Dec. PMID 35572360
- [Background] Kurdahi Badr L, Demerjian T, Daaboul T, Abbas H, Hasan Zeineddine M, Charafeddine L. Preterm infants exhibited less pain during a heel stick when they were played the same music their mothers listened to during pregnancy. Acta Paediatr. 2017 Mar;106(3):438-445. doi: 10.1111/apa.13666. Epub 2016 Dec 13. PMID 27883227